CLINICAL TRIAL: NCT01567436
Title: A Prospective Study of Male Circumcision Using the Shang Ring in Routine Clinical Settings in Kenya & Zambia
Brief Title: A Prospective Field Study: Introducing the Shang Ring in Routine Clinical Settings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); EngenderHealth (Other); Weill Medical College of Cornell University (Other); Kenya National AIDS & STI Control Programme (Other); Ministry of Medical Services, Kenya (Other); University Teaching Hospital, Lusaka, Zambia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10728
Record Dates: First submitted 2012-02-28; First posted 2012-03-30 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Male Circumcision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Shang Ring — The Shang Ring is a sterile device consisting of two concentric medical grade plastic rings: an inner ring with a silicone band and an outer, hinged ring. The inner ring fits inside the outer ring which will lock when snapped together. The Shang Ring comes in multiple sizes. The appropriate size is determined through use of a measuring strip. To ensure that men cannot remove the device prematurely, the locking mechanism must be broken open using a tool that is similar to a scalpel handle. Then, a pair of scissors is used to remove the inner ring, and a bandage or gauze dressing is applied.

SUMMARY:
Male Circumcision (MC) is the only new biomedical method to demonstrate consistent efficacy as an HIV prevention intervention in randomized controlled trials (WHO and UNAIDS, 2007), based on three randomized controlled trials in Kenya, Uganda, and South Africa, that reported a protective effect of about 60%

DETAILED DESCRIPTION:
The World Health Organization, the Joint United Nations Programme on HIV/AIDS (UNAIDS), and other global reproductive health organizations have recognized the highly protective effect of male circumcision to prevent HIV infection in men. Male Circumcision (MC) is the only new biomedical method to demonstrate consistent efficacy as an HIV prevention intervention in randomized controlled trials, based on three randomized controlled trials in Kenya, Uganda, and South Africa, that reported a protective effect of about 60%. Subsequent studies have confirmed the value and persistence of MC's protection against HIV infection, and have demonstrated that MC also reduces the transmission of human papillomavirus.

A wide variety of instruments, devices, and techniques are used around the world for male circumcision. The WHO, UNAIDS and JHPIEGO document entitled Manual for Male Circumcision under Local Anesthesia, includes step-by-step instructions for performing adult male circumcision using three different surgical procedures: the forceps-guided, dorsal slit, and sleeve resection methods. Procedure times for these techniques are approximately 20-30 minutes excluding anesthesia and involve control of unavoidable bleeding and a significant amount of suturing, and can be associated with complications that include hematoma formation, infection, unsatisfactory cosmetic result, lacerations of the penile or scrotal skin and injury to the glans, particularly among inexperienced surgeons. Although training is necessary regardless of method, devices for MC have the potential to reduce both training time and surgical duration because neither hemostasis nor suturing is needed for most devices.

The Shang Ring is an innovative device for adult male circumcision that has been on the Chinese market since 2005. The Shang Ring is manufactured by Wuhu SNNDA Medical Treatment Appliance Technology Co., Ltd (SNNDA).

In the current African setting, only surgical circumcision is available for adults. Devices such as the Shang Ring have the potential to simplify and shorten surgery by eliminating the need for suturing and hemostasis. Data from two small studies in Kenya suggest that the Shang Ring has an acceptable safety profile. A randomized controlled trial was conducted in Kenya and Zambia to provide further data.

Circumcision using the Shang Ring involves a few simple steps. First, a special measuring strip is used to determine which Shang Ring size to use. Following administration of local anesthesia, the inner ring is fitted at the base of the glans penis. Next, the foreskin is everted over the inner ring and the outer ring is secured (locked) over the inner ring, thus encasing the foreskin. The sterile device forms a tight seal. The foreskin is excised and several nicks are made in the foreskin on the underside of the device to prevent formation of a stiff, circumferential scab. Bleeding is minimal and no suturing or hemostasis is required. Finally, the participant returns in seven days for removal of the Shang Ring device. After removal, a bandage is applied to the wound. Men may be given a supply of bandages and told to change the bandaging daily or as needed.

ELIGIBILITY:
Inclusion Criteria:

All men enrolled in this research study must meet the following inclusion criteria:

* Must be aged 18 and 54 years;
* Must be uncircumcised (on examination);
* Must be in good general health;
* Must agree to HIV counseling and testing no more than one week before the procedure;
* Must be free of genital ulcerations or other visible signs of STI (on examination);
* Must be able to understand study procedures and requirements of study participation;
* Must agree to return to the healthcare facility for the full schedule of follow-up visits after his circumcision;
* Must freely consent to participate in the study and sign a written informed consent form;
* Must have a cell phone or access to a cell phone; and,
* Must agree to provide the study staff with an address, phone number, or other locator information while participating in the research study.

Exclusion Criteria:

* A man will be excluded from participation in this research study if he has any of the following exclusion criteria:

  * Has a known allergy or sensitivity to lidocaine or other local anesthesia;
  * Takes a medication that would be a contraindication for elective surgery, such as an anticoagulant or steroid;
  * Has known bleeding/clotting disorder (e.g. hemophilia); or
  * Has an active genital infection, anatomic abnormality or other condition (e.g. severe obesity, diabetes or sickle cell anemia), which in the opinion of the surgeon, prevents the man from undergoing a circumcision as part of this study;
  * Is currently participating in another biomedical study.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 42 days

SECONDARY OUTCOMES:
Acceptability of the Shang Ring Procedure | 42 days
Percentage of men completely healed at 42 days | 42 Days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Goldstein, M.D., Study Chair — Weill Cornell Medical College, NY, USA; Mark A Barone, DVM, MS, Study Chair — EngenderHealth, NY, USA; Philip S Li, MD, Principal Investigator — Weill Cornell Medical College, NY, USA; Richard Lee, MD, Principal Investigator — Weill Cornell Medical College, NY, USA; Paul Perchal, MA, Principal Investigator — EngenderHealth, NY, USA; Jared Mogouche, MD ChB, Principal Investigator — EngenderHealth, Kisumu, Kenya; Quentin Awori, MB ChB, Principal Investigator — EngenderHealth, Homa Bay, Kenya; Raymond Simba, MB ChB MPH, Principal Investigator — Homa Bay District Hospital, Ministry of Health, Homa Bay, Kenya; Nicholas Muraguri, MB ChB MPH, Principal Investigator — National AIDS/STD Control Programme, Nairobi, Kenya; John M Wekesa, MB ChB MMed, Principal Investigator — Ministry of Medical Services, Nairobi, Kenya; Kasonde Bowa, MSc M. Med FRCS FACS FCS, Principal Investigator — University of Zambia; Robert Zulu, MD, Principal Investigator — University Teaching Hospital, Lusaka, Zambia
Locations (2):
- Homa Bay District Hospital male circumcision clinic, Homa Bay, Nyanza, Kenya
- Society for Family Planning Clinic, Lusaka, Lusaka Province, Zambia

REFERENCES:
- [Derived] Barone MA, Li PS, Zulu R, Awori QD, Agot K, Combes S, Simba RO, Lee RK, Hart C, Lai JJ, Zyambo Z, Goldstein M, Feldblum PJ, Sokal DC. Men's Understanding of and Experiences During the Postcircumcision Abstinence Period: Results From a Field Study of ShangRing Circumcision During Routine Clinical Services in Kenya and Zambia. J Acquir Immune Defic Syndr. 2016 Jun 1;72 Suppl 1(Suppl 1):S18-23. doi: 10.1097/QAI.0000000000000704. PMID 27331585
- [Derived] Feldblum PJ, Okech J, Ochieng R, Hart C, Kiyuka G, Lai JJ, Veena V. Longer-Term Follow-Up of Kenyan Men Circumcised Using the ShangRing Device. PLoS One. 2015 Sep 14;10(9):e0137510. doi: 10.1371/journal.pone.0137510. eCollection 2015. PMID 26367141